CLINICAL TRIAL: NCT05263700
Title: FAPI-CUP - Evaluating FAPI as a Novel Radiopharmaceutical Targeting Cancer-associated Fibroblasts for the Diagnosis of Patients With Cancer of Unknown Primary
Brief Title: FAPI-CUP- Evaluating FAPI as a Novel Radiopharmaceutical for Cancer of Unknown Primary
Acronym: FAPI-CUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PMC71838
Record Dates: First submitted 2022-02-15; First posted 2022-03-03 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cancer of Unknown Primary Site
Keywords: FAPI; PET/CT; CUP; FAPI-46
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — FAPI-46

STUDY DESIGN:
Intervention Model Description: This is a prospective single arm cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-PET/CT (Experimental): Patients receive 68Ga-FAPI IV then undergo PET/CT.
  Interventions: Drug: 68Ga-FAPi-46; Procedure: PET/CT imaging

INTERVENTIONS:
Drug: 68Ga-FAPi-46 — FAPI-46 is a small molecular radiopharmaceutical that binds to the fibroblast activated protein on cancer associated fibroblasts. Gallium-68 (68Ga) is a positron-emitting isotope with a half-life of 68 minutes.
Procedure: PET/CT imaging — PET with the investigational tracer 68Ga-FAPI-46 with accompanying low-dose CT for anatomical localisation

SUMMARY:
This is a prospective single arm cohort study designed to evaluate the diagnostic ability of 68Ga-FAPI-PET/CT scan in determining likely tissue of origin in Cancer of Unknown Primary (CUP) patients not identified by standard of care. Patients with CUP will be either treatment naïve or starting second-line treatment.

DETAILED DESCRIPTION:
Cancers of unknown primary (CUP) account for 3-5% of all malignancies. The prognosis of patients diagnosed with CUP is poor, with a median overall survival of 9-12 months. Despite improvements in conventional diagnostic processes, the tissue of origin (ToO) is identified in <30% of CUP patients. PET/CT is increasingly used to determine the ToO, with the most commonly used PET radiotracer being the glucose analogue fluorine-18 fluorodeoxyglucose (FDG). Although PET/CT can change CUP patient management and identify primary sites, FDG has limited sensitivity for detecting some cancers, such as CUP. It has been reported that fibroblast activation protein (FAP) is highly expressed in some tumours, including CUP. 68Ga-FAPI (experimental drug) is a radiotracer that can specifically bind to FAP, and may enable the primary cancer site to be viewed using PET imaging. It is hypothesised that the use of 68Ga-FAPI-PET/CT will increase likely ToO diagnosis from 30% with current standard of care to 60%.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent
2. Participants aged 18 years or over at screening
3. Diagnosed with CUP based on a diagnostic work-up, including, but not limited to; a detailed clinical assessment; a CT scan of the chest/abdomen, and pelvis; pathological review of tumour tissue; and other appropriate tests as per the Cancer Council Optimal Care Pathway guidelines
4. Has not commenced current line of systemic treatment
5. Eastern Cooperative Oncology Group performance status 0 - 2
6. Life expectancy greater than 3 months
7. Adequate hematologic and organ function to commence systemic treatment, defined by the following laboratory results:

   1. Haemoglobin ≥ 90g/L
   2. Absolute neutrophil count ≥1.5 x 109/L
   3. Platelet count ≥ 100 x 109/L
   4. Creatinine clearance ≥ 30mL/min
   5. Serum bilirubin ≤ 1.5 x upper limit of normal (ULN); patients with known Gilbert's disease may have a bilirubin ≥ 3.0 x ULN
   6. Aspartate transaminase (AST) or alanine transaminase (ALT) ≤2 x ULN (or ≤ 5 x ULN in the presence of liver metastases)
8. Willing and able to comply with all study requirements, including all treatment and required assessments including follow-up procedures, in the investigator's judgment

Exclusion Criteria:

1. Uncontrolled medical or psychological conditions that may prevent commencement of systemic treatment.
2. Major surgical procedure within 6 weeks prior to study registration or active infection requiring systemic treatment

   a. Placement of vascular access devices is not considered major surgery.
3. Concurrent illness, including severe infection that may jeopardise the ability of the participant to undergo procedures outlined in this protocol with reasonable safety
4. Prior cancer diagnosis with the exception of:

   1. Malignancy treated with curative intent and with no known active disease ≥ 3years and of low potential risk of recurrence
   2. Adequately treated basal cell or squamous cell skin carcinoma or non-invasive melanoma
   3. Adequately treated non-muscle invasive bladder cancer (Tis, Ta and low grade T1 tumours)
   4. Adequately treated carcinoma in situ without evidence of disease
   5. Cancer subjects with incidental histologic findings of prostate cancer that, in the opinion of the Investigator, is not deemed to require active therapy (e.g., incidental prostate cancer identified following cystoprostatectomy that is tumour/node/metastasis stage ≤ pT2N0)
5. Greater than one prior line of systemic treatment
6. Known allergy or reaction to 18F or 68Ga tracer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-02-22 (Estimated); Study Completion 2024-02-22 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients in which a likely tissue of origin is identified using 68Ga-FAPI-PET/CT | 12 months
  The proportion of patients in which 68Ga-FAPI-PET/CT identifies a likely Tissue of Origin (ToO) beyond that identified by standard of care (SoC) testing.

SECONDARY OUTCOMES:
Maximum Standard Uptake Value measured on 68Ga-FAPI-PET/CT | 12 months
  The average SUVmax of the 5 most intense lesions measured on 68Ga-FAPI-PET/CT based on the best overall response rate assessed via RECIST after commencement of systemic therapy.
The proportion of patients in which the choice of treatment is changed after the 68Ga-FAPI-PET/CT | 12 months
  The change in patient management/treatment pre- and post- 68Ga-FAPI-PET/CT.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Bendigo Health, Bendigo, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - South West Healthcare, Warrnambool, Victoria

IPD SHARING:
Plan to Share IPD: No